CLINICAL TRIAL: NCT03187314
Title: Phase II Study of Radiation Therapy With Anti-PD-1 Antibody SHR-1210 in Treating Patients With Unresectable Esophageal Cancer
Brief Title: Combination of Radiation Therapy and Anti-PD-1 Antibody SHR-1210 in Treating Patients With Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shixiu Wu, Professor, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH08
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Esophageal Neoplasms; Esophageal Diseases; Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Radiation; Anti-PD-1 Antibody
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases; Esophageal Squamous Cell Carcinoma | interventions — Radiation; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Radiation to 60 Gy, 5 x per week, for 6 weeks. Radiation begun the day after the first dose of SHR-1210. SHR-1210 (200mg fixed dose every 2 weeks for 5 cycles) will be administered as an intravenous infusion over 60 minutes.
  Interventions: Drug: Radiation; Drug: SHR-1210

INTERVENTIONS:
Drug: Radiation — RT to 60 Gy, 5 x per week，for 6 weeks. Radiation begun the day after the first dose of SHR-1210
Drug: SHR-1210 — SHR-1210 (200mg fixed dose every 2 weeks for 5 cycles) will be administered as an intravenous infusion over 60 minutes.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of radiation therapy combined with anti-PD-1 antibody SHR-1210 in patients with esophageal cancer

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or femal.
2. Histologically or cytologically confirmed Squamous Cell Carcinoma of the Esophagus, locally advanced, unresectable disease.
3. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
4. Can provide either a newly obtained or archival tumor tissue sample.
5. ECOG 0-1.
6. Life expectancy of greater than 12 weeks.
7. Adequate organ function.
8. Female: child bearing potential, a negative urine or serum pregnancy test result within 72 h before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study through 3 months after the last dose of SHR-1210.
9. Patient has given written informed consent.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. Complete obstruction of the esophagus, or patients who have the potential to develop perforation
3. Other malignancy within 5 years prior to entry into the study, expect for curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers.
4. Known central nervous system (CNS) metastases.
5. Subjects with any active autoimmune disease or history of autoimmune disease.
6. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
7. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
8. History of Interstitial Pneumonia or active non-infectious pneumonitis.
9. Known Human Immunodeficiency Virus (HIV) infection、active Hepatitis B or Hepatitis C.
10. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agent.
11. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR-1210 formulation.
12. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treament. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalen for replacement therapy.
13. Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent.
14. Received a live vaccine within 4 weeks of the first dose of study medication.
15. Pregnancy or breast feeding.
16. Decision of unsuitableness by principal investigator or physician-in-charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 4-8 weeks
  ORR was evaluated 4-8 weeks after completion of RT and was recorded according to RECIST, version 1.1.

SECONDARY OUTCOMES:
Treatment-emergent adverse events | year 0 - year 1
  Incidence of treatment-emergent adverse events would be assessed based on the common toxicity criteria for adverse events version 4.0 (CTCAE v4.0) and EORTC criterion.
Local-regional free survival (LRFS) | year 0 - year 3
  LRFS was calculated from the date of treatment initiation to the date of documented failure.
Overall survival | year 0 - year 3
  OS was determined as the time (in months) between the first day of therapy and the last follow-up or the date of death.
Health-related quality of life (HRQoL) | From baseline to one year after RT.
  HRQoL measured by standardized EORTC questionaires (EORTC QLQ-C30)
Health-related quality of life (HRQoL) | From baseline to one year after RT.
  HRQoL measured by standardized EORTC questionaires (EORTC QLQ-OES18)

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided